CLINICAL TRIAL: NCT04665752
Title: Ocular Findings and Viral Persistence in Ocular Fluids in COVID-19 Survivors, a Natural History, Observational Study
Brief Title: Ocular Findings and Viral Persistence in Ocular Fluids in COVID-19 Survivors
Status: Terminated | Type: Observational
Why Stopped: Slow/Insufficient accrual
Sponsor: National Eye Institute (NEI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 10000078; 000078-EI
Record Dates: First submitted 2020-12-11; First posted 2020-12-14 (Actual); Last update posted 2022-10-06 (Actual); Status verified 2022-10

CONDITIONS: COVID-19
Keywords: Images; Natural History
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Affected Participants: Participants previously diagnosed with COVID-19.

SUMMARY:
Background:

Some people who have had COVID-19 experience changes in the eye. Sometimes these changes are subtle and may not affect vision. Researchers want to learn how many people experience these eye changes and where in the eye they occur to better understand the outcomes of COVID-19 and its treatments.

Objective:

To examine possible changes in the eye that might have occurred as a result of COVID-19.

Eligibility:

Adults age 18 and older who were diagnosed with COVID-19 and recovered.

Design:

Participants will be screened with a medical history and physical exam. They will have blood tests.

Participants will have an eye exam. Their pupils will be dilated with eye drops. Eye pressure and movements will be measured.

Participants will have optical coherence tomography. Pictures will be taken of the retina and the inside of the eyes.

Participants may have fluorescein angiography and indocyanine green angiography. They will be given a dye through an intravenous line. The dye will travel up to the blood vessels in their eyes. Pictures will be taken of the dye as it flows through the blood vessels.

Participants may have electroretinography to test the retina. They will sit in the dark with their eyes patched for 30 minutes. Then they will watch flashing lights while wearing contact lenses that sense signals from the retina.

Participants may have adaptive optics-assisted imaging. They will look at a specific location while images are taken of the retina.

During the study, participants will have blood drawn through a needle in their arm. Fluid or tissue from the eye may be obtained if participants have a medically needed procedure.

Participation will last for 12 months.

DETAILED DESCRIPTION:
Study Description:

The objective of this study is to understand the rate and extent of ocular involvement in COVID-19 patients and whether SARS-COV-2 can be detected in ocular fluids or tissue in convalescent phase.

Objectives:

Primary Objective: To investigate if COVID survivors show signs of anterior or posterior segment inflammation or other retinochoroidal changes after recovery.

Secondary Objectives:

To investigate if SARS-Cov-2 can be detected in the ocular fluids or tissues of survivors among patients who undergo medically indicated ocular surgery or diagnostic procedures.

Exploratory Objective: To investigate whether the use of chloroquine/Hydroxychloroquine for treatment of COVID-19 is associated with ocular changes.

Endpoints:

Primary Endpoint: Percentage of patients with Ocular exam abnormalities such as conjunctival/corneal, anterior segment, choroidal, retinal lesions and subclinical findings on OCT, FA and ICG

Secondary Endpoints:

Correlation of ocular findings with COVID severity (by history)

Proportion of patients with +SARS-COV-2 PCR in ocular fluid/tissues among COVID-19 survivors and correlation to clinical characteristics and IgG levels

Study Population:

Up to 150 COVID-19 survivors will be recruited.

Description of Sites/Facilities Enrolling Participants:

This protocol will enroll participants at the NIH CC. De-identified samples may be received from the New York Medical Center.

Study Duration:

2 years

Participant Duration:

The participants will be asked to come to the NIH CC for one visit. A select subgroup of up to 75 participants with positive findings may be asked to return within 12 months from their initial visit.

ELIGIBILITY:
* INCLUSION CRITERIA:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

1. Stated willingness to comply with all study procedures and availability for the duration of the study
2. Male or female, aged 18 or older.
3. History of positive PCR or positive IgG for SARS-CoV-2 cases and if known history of COVID-19 infection, at least 30 days passed since a positive PCR for SARS-COV-2 and have been asymptomatic for at least 10 days.
4. Willing to undergo study required testing and blood draw.
5. Willing to have blood samples stored for future research.

EXCLUSION CRITERIA:

An individual who meets any of the following criteria will be excluded from participation in this study:

1. Current symptoms consistent with COVID-19 infection.
2. Any condition or event that, in the PI s opinion, may substantially increase the risk associated with study participation or compromise the study's scientific objectives. Conditions that exclude a subject are considered to be unlikely, but an example would include having an acute respiratory infection or recent exposure that would make it unsafe to perform study procedures or obtain blood samples.
3. Pregnant and decisionally impaired individuals will be excluded from participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants diagnosed with COVID-19 and at least 30 days symptom-free.
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2021-02-02 (Actual); Primary Completion 2022-01-28 (Actual); Study Completion 2022-01-28 (Actual)

PRIMARY OUTCOMES:
Percentage of participants | Over the study duration
  Percentage of participants with ocular exam abnormalities, such as conjunctival/corneal anterior segment, choroidal, retinal lesions and subclinical findings on OCT, FA, and ICG.

SECONDARY OUTCOMES:
Correlation of findings | Over the study duration
  Correlation of ocular findings with COVID severity
Proportion of patients | Over the study duration
  Proportion of patients with +SARS-COV-2 PCR in ocular fluid/tissues among COVID-19 survivors and correlation to clinical characteristics and IgG levels.

CONTACTS AND LOCATIONS:
Overall Officials: Shilpa M Kodati, M.D., Principal Investigator — National Eye Institute (NEI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_000078-EI.html